CLINICAL TRIAL: NCT06369428
Title: Non-interventional Register-based Study to Analyze Patient Characteristics, Treatment Patterns and Healthcare Resource Utilization in Adult Patients With Metastatic Melanoma
Brief Title: Patient Characteristics, Treatment Patterns, and Healthcare Resource Utilization of Metastatic Melanoma Patients
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CDRB436BFI02
Record Dates: First submitted 2024-04-11; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Distant Metastasis Cohort: Adult patients diagnosed with stage 4 (distant) metastatic melanoma between 2014 and 2021.
- Regional Metastasis Cohort: Adult patients diagnosed with stage 3 (regional) metastatic melanoma between 2014 and 2021.

SUMMARY:
This was a retrospective, non-interventional, registry study based on secondary electronic medical record (EMR) data collected in Helsinki and Uusimaa hospital district (HUS data lake), hospital district of Southwest Finland (VSSHP data lake) and Pirkanmaa hospital district (PSHP data lake) as a part of their routine clinical practice. Social Insurance Institution of Finland (SII; reimbursed drug purchases) was utilized in this study to complement the medication data. The metastatic melanoma patients were stratified by first-line treatment and by hospital district.

ELIGIBILITY:
Inclusion criteria

* Patients diagnosed with metastatic melanoma (C43) during 01 January 2014 and 31 December 2021.
* Adult (18 years or older) at the time of diagnosis of metastatic melanoma.
* Resident in the corresponding hospital district(s) at the time of diagnosis of metastatic melanoma.

Exclusion criteria

* Metastasis recorded prior to 01 January 2014 (i.e. prevalent case).
* Record of any other cancer (The International Classification of Diseases, 10th Revision [ICD-10] diagnosis code starting with C, excluding C43, C77, C78, and C79) as last cancer diagnosis before metastasis.
* Participated in COBRA (vemurafenib, temozolomide, lomustine, vincristine) trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 1795 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Mean Age-standardized Annual Incidence of Metastatic Melanoma in 2014-2021 | Up to approximately 7 years
Point Prevalence per 100,000 Population | Up to approximately 7 years
  Point prevalence was defined as the number of metastatic melanoma patients alive at the end of 2021 divided by the total of hospital districts of Helsinki and Uusimaa hospital district (HUS), Pirkanmaa hospital district (PSHP), and Hospital district of Southwest Finland (VSSHP).
Mean Age of Patients at Index Date per Hospital District | Index date, defined as date of metastasis diagnosis
Mean Length of Follow-up at Index Date per Hospital District | Index date, defined as date of metastasis diagnosis
Gender at Index Date per Hospital District | Index date, defined as date of metastasis diagnosis
Number of Patients with Lactate Dehydrogenase (LDH) Levels Less than the Upper Limit of Normal (ULN) at Index Date per Hospital District | Index date, defined as date of metastasis diagnosis
Number of Patients with LDH Levels Between the ULN and 1.5 Times ULN at Index Date per Hospital District | Index date, defined as date of metastasis diagnosis
Number of Patients with LDH Levels Greater than 1.5 Times ULN at Index Date per Hospital District | Index date, defined as date of metastasis diagnosis
Number of Patients with Positive Proto-oncogene B-Raf (BRAF) Status at Index Date per Hospital District | Index date, defined as date of metastasis diagnosis
Number of Patients with Negative BRAF Status at Index Date per Hospital District | Index date, defined as date of metastasis diagnosis
Number of Patients by Charlson Comorbidity Index (CCI) Score Category at Index Date per Hospital District | Index date, defined as date of metastasis diagnosis
  CCI predicts the ten-year mortality for a patient who may have a range of comorbid conditions. Comorbidity was assessed using the CCI, categorized as low (0-1) and high (≥2).
Number of Patients by Number of Metastatic Organs at Index Date per Hospital District | Index date, defined as date of metastasis diagnosis
Number of Patients by Location of Metastases at Index Date per Hospital District | Index date, defined as date of metastasis diagnosis
  Locations of metastatic sites at study entry:
  * lymph node
  * lung
  * skin/subcutaneous
  * liver
  * brain
  * bone
  * kidney
  * peritoneum/peritoneal cavity
  * spleen
  * pancreas
  * intestine
Number of Patients by Tumor, Nodes, and Metastasis (TNM) Stage per Hospital District | Index date, defined as date of metastasis diagnosis
Number of Patients by Most Prevalent (greater than 5%) Baseline Comorbidities per First-line Medication | 5 years prior to index date, where index date was defined as date of metastasis diagnosis

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 7 years
  Overall survival was defined as the time from the index date until death or to end of study follow-up. Index date was defined as date of metastasis diagnosis.
Time to Next Treatment (TTNT) of the First-line (1L) by Type of Treatment | Up to approximately 7 years
  TTNT was defined as the time from initiation of a treatment line until the initiation of the next treatment line, death, or end of study follow-up.
Duration of Treatment (DoT) | Up to approximately 7 years
  DoT was defined as the time from initiation of a treatment line until the end of treatment, death, or end of study follow-up.
Mean Age at Index Date per First-line (1L) Medication | Index date, defined as date of metastasis diagnosis
Length of Follow-up at Index Date per 1L Medication | Index date, defined as date of metastasis diagnosis
Time to Treatment at Index Date per 1L Medication | Index date, defined as date of metastasis diagnosis
Gender at Index Date per 1L Medication | Index date, defined as date of metastasis diagnosis
Number of Patients with Lactate Dehydrogenase (LDH) Levels Less than the Upper Limit of Normal (ULN) at Index Date per 1L Medication | Index date, defined as date of metastasis diagnosis
Number of Patients with LDH Levels Between the ULN and 1.5 Times ULN at Index Date per 1L Medication | Index date, defined as date of metastasis diagnosis
Number of Patients with LDH Levels Greater than 1.5 Times ULN at Index Date per 1L Medication | Index date, defined as date of metastasis diagnosis
Number of Patients with Positive Proto-oncogene B-Raf (BRAF) Status at Index Date per 1L Medication | Index date, defined as date of metastasis diagnosis
Number of Patients with Negative BRAF Status at Index Date per 1L Medication | Index date, defined as date of metastasis diagnosis
Number of Patients by Charlson Comorbidity Index (CCI) Score Category at Index Date per 1L Medication | Index date, defined as date of metastasis diagnosis
  CCI predicts the ten-year mortality for a patient who may have a range of comorbid conditions. Comorbidity was assessed using the CCI, categorized as low (0-1) and high (≥2).
Number of Patients by Number of Metastatic Organs at Index Date per 1L Medication | Index date, defined as date of metastasis diagnosis
Number of Patients by Location of Metastases at Index Date per 1L Medication | Index date, defined as date of metastasis diagnosis
  Locations of metastatic sites at study entry:
  * lymph node
  * lung
  * skin/subcutaneous
  * liver
  * brain
  * bone
  * kidney
  * peritoneum/peritoneal cavity
  * spleen
  * pancreas
  * intestine
Number of Patients by Tumor, Nodes, and Metastasis (TNM) Stage per 1L Medication | Index date, defined as date of metastasis diagnosis
Number of Patients that Received Radiotherapy During 1L Treatment | Index date, defined as date of metastasis diagnosis
Number of Patients Switched from Immuno-oncology (IO) 1L Treatment to Targeted Therapy (TT) Second-line (2L) Treatment | Up to approximately 7 years
Number of Patients Switched from IO 1L Treatment to Chemotherapy (Chemo) 2L Treatment | Up to approximately 7 years
Number of Patients Switched from TT 1L Treatment to IO 2L Treatment | Up to approximately 7 years
Number of Patients Switched from TT 1L Treatment to Chemo 2L Treatment | Up to approximately 7 years
Number of Patients Switched from Chemo 1L Treatment to IO 2L Treatment | Up to approximately 7 years
Number of Patients Switched from Chemo 1L Treatment to TT 2L Treatment | Up to approximately 7 years
Number of Patients Switched from IO 2L Treatment to TT Third-line (3L) Treatment | Up to approximately 7 years
Number of Patients Switched from IO 2L Treatment to Chemo 3L Treatment | Up to approximately 7 years
Number of Patients Switched from TT 2L Treatment to IO 3L Treatment | Up to approximately 7 years
Number of Patients Switched from TT 2L Treatment to Chemo 3L Treatment | Up to approximately 7 years
Number of Patients Switched from Chemo 2L Treatment to IO 3L Treatment | Up to approximately 7 years
Number of Patients Switched from Chemo 2L Treatment to TT 3L Treatment | Up to approximately 7 years
Number of Healthcare Contacts and Associated Costs per Patient Year | Up to approximately 7 years
  Costs of outpatient visits, hospitalizations, and emergency room (ER) visits were estimated using unit costs and thus contain an average cost of performed procedures and operations, analyzed laboratory tests, and given medications (i.e. hospital inpatient medications) during the healthcare contact.
Number of Healthcare Contacts and Associated Costs per Patient | Up to approximately 7 years
  Costs of outpatient visits, hospitalizations, and emergency room (ER) visits were estimated using unit costs and thus contain an average cost of performed procedures and operations, analyzed laboratory tests, and given medications (i.e. hospital inpatient medications) during the healthcare contact.
Number of Healthcare Contacts and Associated Total Costs | Up to approximately 7 years
  Costs of outpatient visits, hospitalizations, and emergency room (ER) visits were estimated using unit costs and thus contain an average cost of performed procedures and operations, analyzed laboratory tests, and given medications (i.e. hospital inpatient medications) during the healthcare contact.

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis, Basel, Switzerland